CLINICAL TRIAL: NCT03061227
Title: Metabolic and Central Nervous System Characterisation of the Phenotype of Non-suppressed (Rising) Glucagon After Glucose Challenge
Brief Title: Characterization of Metabolic and Brain Effects of Rising Glucagon During an Oral Glucose Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 529_2016BO1
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Metabolic Syndrome; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous glucagon (Active Comparator): Low-dose glucagon infusion (0.5 pmol/min/kg body weight) over 150 minutes during a standardized 75 g oral glucose tolerance test
  Interventions: Drug: Intravenous glucagon
- Intravenous saline (Placebo Comparator): Saline infusion over 150 minutes during a standardized 75 g oral glucose tolerance test
  Interventions: Drug: Intravenous saline

INTERVENTIONS:
Drug: Intravenous glucagon — Randomized application of glucagon or saline during oral glucose tolerance test
  Arms: Intravenous glucagon
Drug: Intravenous saline — Randomized application of glucagon or saline during oral glucose tolerance test
  Arms: Intravenous saline

SUMMARY:
The investigators previously characterized a phenotype with non-suppressed glucagon at 120 minutes after standardized oral glucose load. This phenotype is associated with healthy metabolic traits such as lower BMI, higher insulin sensitivity and lower liver fat content. Glucagon is a pleiotropic hormone that, besides its main action on increasing endogenous glucose production, also reduces appetite and increases basal energy expenditure. The aims of this study are to i. detect functional differences in the appetite-related central nervous system (CNS) areas between the suppressed and non-suppressed glucagon phenotype ii. mimick the non-suppressed glucagon phenotype in those participants who suppress glucagon by administering a very-low-dose glucagon infusion and retest them.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5- 29.9 kg/m2
* written informed consent

Exclusion Criteria:

* Current

  1. febrile infection with temperatures> 38.5 ° C in the last 14 days
  2. Blood donation within the last 12 weeks Pre-study Inclusion
* Chronic diseases:

  1. Diabetes mellitus
  2. Known liver diseases (hepatitisB/C, hemochromatosis, NASH)
  3. Chronic inflammatory diseases (rheumatoid arthritis, Crohn's disease, ulcerative colitis) chronic renal insufficiency
  4. Cancer (known malignant disease)
  5. psychiatric diagnoses (bipolar disorder, schizophrenia, psychoses, depression, agoraphobia)
  6. Persons with non-removable metal parts, e.g:

     * pacemaker
     * artificial heart valves
     * metal prostheses
     * implanted magnetic metal parts (screws, plates of operations)
     * spiral
     * metal slivers / garnet splinters
     * fixed braces
     * Acupuncture needle
     * Insulin pump
     * totally implantable venous access device (port)
     * tattoos, metallic eye shadows
  7. Persons with impaired sensitivity and / or increased sensitivity to heating of the body
  8. Medical history of venous thromboembolism
  9. alcohol consumption of more than 50g / day
  10. In physical examination:

      blood pressure > 160/100 mmHg pathologic cardiac murmurs (diastolic or systolic louder than 2/6)
  11. in the blood test: fasting glucose ≥ 125 mg/dl or HbA1c ≥ 6.5% AST or ALT> 2.5x upper limit of the reference range (> 125 U/l) Hb <12 g/dl C reactive protein (CRP) > 5 mg / dL or leukocytes> 15000/μl

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Brain activity | change from baseline to 120 minutes after oral glucose challenge
  Resting-state brain activity assessed by fMRI

SECONDARY OUTCOMES:
Hunger rating | before and 150 minutes after oral glucose challenge and start of glucagon/saline infusion
  On visual analogue scale
Brain response to food cues | before, 30 minutes and 120 minutes after oral glucose challenge and start of glucagon/saline infusion
  Assessed by functional magnetic resonance imaging (fMRI)
Glucose tolerance | 0-120 minutes
  Assessed by 75 g oral glucose tolerance test
Insulin sensitivity | 0-120 minutes
  Assessed during 75 g oral glucose tolerance test
Basal energy expenditure | 150 minutes after oral glucose challenge
  Assessed by indirect calorimetry
Change in hormone levels | 0-150 minutes
  Change in adrenocorticotropic hormone (ACTH), growth hormone (GH), thyroid-stimulating hormone (TSH), luteinizing hormone (LH), follicle stimulating hormone (FSH), fibroblast growth factor 21(FGF-21) after oral glucose challenge and start of glucagon/saline infusion.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No